CLINICAL TRIAL: NCT02978547
Title: The Effects of Neoadjuvant Metformin on Tumour Cell Proliferation and Tumour Progression in Pancreatic Ductal Adenocarcinoma
Acronym: Metformin 001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Pancreatic Cancer Canada (Other); BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H16-02566
Record Dates: First submitted 2016-11-02; First posted 2016-12-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma
Keywords: Resectable pancreatic ductal adenocarcinoma; PDAC; Metformin
MeSH Terms: interventions — Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): All patients will receive metformin 500 mg per oral twice daily with food for at least 7 days, until 2 days prior to surgery. Metformin therapy should be discontinued 2 days before surgery to reduce the risk of lactic acidosis associated with fasting.
  Interventions: Drug: Metformin Hydrochloride 500Mg Tablet

INTERVENTIONS:
Drug: Metformin Hydrochloride 500Mg Tablet — In the event of any grade 2 toxicities (with the exception of hyperglycemia), metformin will be withheld until improvement to ≤ grade 1, then restarted at a dose of 500 mg daily. In the event of grade ≥ 3 toxicities related to metformin, treatment will be discontinued. Metformin therapy will also be discontinued if serum lactate levels are above normal values.

SUMMARY:
This is a single arm, non-randomized phase II study of neoadjuvant metformin in resectable PDAC. Twenty patients will be enrolled and treated with metformin 500 mg BD for a minimum of 7 days, until 2 days prior to surgery. Patients will undergo laboratory investigations at baseline, prior to surgery and 4-10 weeks after surgery. Patients eligible for and consented to the optional MRI substudy will undergo diffusion-weighted MRI 1 to 14 days before surgery.

At surgery, resected tumour and normal tissue will be collected and banked. FFPE specimens will be used for sectioning, histological analysis and IHC for Ki67 (cell proliferation marker), pAMPK, ACC targets, p53 and mTOR targets, apoptotic markers (Bax, Bcl-2, caspases 3, 8 and 9). Fresh frozen tumour and matched normal tissue samples will be used for western blot analysis of insulin and IGF receptors, total and activated ERK and Akt, and RNAseq analysis. Pre-metformin biopsy samples will be retrieved for molecular analysis.

Fasting blood samples at baseline and before surgery will be analyzed for glucose and insulin levels. Plasma and whole blood will also be processed and banked for circulating tumour DNA analysis. Urine samples will be sent for metabolomic profiling.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years on the day of study consent
* Pathologic diagnosis of PDAC where 2 pre-treatment core biopsy samples are available for analysis. Patients with suspected PDAC without a pathologic diagnosis must undergo confirmatory biopsy under endoscopic ultrasound guidance.
* Resectable disease based on standard imaging criteria
* Surgery planned ≥ 2 weeks after study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematologic, renal, and hepatic function as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:

  * Total bilirubin < 1.5 times the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 times the ULN
  * Lipase < 1.5 times the ULN
  * Serum creatinine < 1.5 times the ULN
  * Glomerular filtration rate > 30 mL/min/1.73 m2 according to the modified diet in renal disease abbreviated formula
  * International normalized ratio (INR) or prothrombin time (PT; PT-INR) and partial thromboplastin time (PTT) < 1.5 times the ULN
  * Platelet count > 100000 /mm3, hemoglobin (> 9 g/dL, absolute neutrophil count > 1500/mm3.
* Baseline fasting glucose <13.9 mmol/L
* No prior chemotherapy or radiotherapy for PDAC
* Serum lactate levels within normal range assessed within 7 days prior to the initiation of study treatment

MRI sub-study:

* Signed informed consent for the optional MRI substudy
* No contraindications to MRI

Exclusion Criteria:

* Presence of locally unresectable disease or distant metastases
* Treatment with metformin or any other anti-hyperglycemic agent within the previous 6 months
* Known allergy or contraindication to metformin
* Not fit for surgery
* Planned for, or received, neoadjuvant treatment of any type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The effect of neoadjuvant metformin treatment on tumour cell proliferation in PDAC tumours | 6 months
  Assessment of Ki-67 fraction as assessed by IHC of pre- and post-metformin tumour samples.

SECONDARY OUTCOMES:
R0 resection rates in patients undergoing curative PDAC resection | 6 months
  Proportion of patients with R0 resections.
The effect of metformin on glucose and insulin metabolism as assessed by serum marker, fasting GGT (mmol/L) | 6 months
  The marker of glucose and insulin metabolism will be reported with pre- and post-metformin values compared.
The effect of metformin on glucose and insulin metabolism as assessed by serum marker, fasting glucose (mmol/L) | 6 months
  The marker of glucose and insulin metabolism will be reported with pre- and post-metformin values compared.
The effect of metformin on glucose and insulin metabolism as assessed by serum marker, fasting insulin (mU/L) | 6 months
  The marker of glucose and insulin metabolism will be reported with pre- and post-metformin values compared.
The effect of metformin on glucose and insulin metabolism as assessed by serum marker, HOMA index | 6 months
  HOMA index is calculated from serum glucose and insulin. The marker of glucose and insulin metabolism will be reported with pre- and post-metformin values compared.
The effect of metformin on glucose and insulin metabolism as assessed by clinical marker, weight (kg) | 6 months
  The clinical marker will be reported with pre- and post-metformin values compared.
The effect of metformin on metabolomic profile of pre- and post-metformin samples | 6 months
  Serum and urine metabolomic profile.
  Comparison of metabolite levels in pre-and post-metformin samples.
Transcriptome sequencing (RNAseq) of pre- and post-treatment tumour samples. | 6 months
  To investigate the molecular signatures associated with metformin response
  Comparison of gene expression in pre-metformin biopsy samples and post-metformin resected tumour samples. Expression of altered genes to be validated by IHC in tumour sections.
Plasma ctDNA, measured as percentage of mutant to total DNA fragments in plasma | 6 months
  To assess the presence of ctDNA in resectable PDAC, and dynamic changes following treatment with metformin and surgical resection
  Proportion of patients with detectable plasma ctDNA at baseline. Comparison of values pre- and post-metformin and 4-10 weeks after surgery.
Correlation between imaging and pathologic parameters | 6 months
  To explore the correlation between apparent diffusion coefficient (ADC) on MRI and pathologic findings.
  ADC values will be individually compared to tumour differentiation and Ki-67 fraction on pathologic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2015. Toronto, ON: Canadian Cancer Society. 2015.
- [Background] Garcea G, Dennison AR, Pattenden CJ, Neal CP, Sutton CD, Berry DP. Survival following curative resection for pancreatic ductal adenocarcinoma. A systematic review of the literature. JOP. 2008 Mar 8;9(2):99-132. PMID 18326920
- [Background] AJCC Cancer Staging Manual. 7th ed. New York: Springer-Verlag; 2010.
- [Background] Callery MP, Chang KJ, Fishman EK, Talamonti MS, William Traverso L, Linehan DC. Pretreatment assessment of resectable and borderline resectable pancreatic cancer: expert consensus statement. Ann Surg Oncol. 2009 Jul;16(7):1727-33. doi: 10.1245/s10434-009-0408-6. Epub 2009 Apr 24. No abstract available. PMID 19396496
- [Background] Gillen S, Schuster T, Meyer Zum Buschenfelde C, Friess H, Kleeff J. Preoperative/neoadjuvant therapy in pancreatic cancer: a systematic review and meta-analysis of response and resection percentages. PLoS Med. 2010 Apr 20;7(4):e1000267. doi: 10.1371/journal.pmed.1000267. PMID 20422030
- [Background] Palmer DH, Stocken DD, Hewitt H, Markham CE, Hassan AB, Johnson PJ, Buckels JA, Bramhall SR. A randomized phase 2 trial of neoadjuvant chemotherapy in resectable pancreatic cancer: gemcitabine alone versus gemcitabine combined with cisplatin. Ann Surg Oncol. 2007 Jul;14(7):2088-96. doi: 10.1245/s10434-007-9384-x. Epub 2007 Apr 24. PMID 17453298
- [Background] Landry J, Catalano PJ, Staley C, Harris W, Hoffman J, Talamonti M, Xu N, Cooper H, Benson AB 3rd. Randomized phase II study of gemcitabine plus radiotherapy versus gemcitabine, 5-fluorouracil, and cisplatin followed by radiotherapy and 5-fluorouracil for patients with locally advanced, potentially resectable pancreatic adenocarcinoma. J Surg Oncol. 2010 Jun 1;101(7):587-92. doi: 10.1002/jso.21527. PMID 20461765
- [Background] Ben Sahra I, Le Marchand-Brustel Y, Tanti JF, Bost F. Metformin in cancer therapy: a new perspective for an old antidiabetic drug? Mol Cancer Ther. 2010 May;9(5):1092-9. doi: 10.1158/1535-7163.MCT-09-1186. Epub 2010 May 4. PMID 20442309
- [Background] Zhang P, Li H, Tan X, Chen L, Wang S. Association of metformin use with cancer incidence and mortality: a meta-analysis. Cancer Epidemiol. 2013 Jun;37(3):207-18. doi: 10.1016/j.canep.2012.12.009. Epub 2013 Jan 24. PMID 23352629
- [Background] Kourelis TV, Siegel RD. Metformin and cancer: new applications for an old drug. Med Oncol. 2012 Jun;29(2):1314-27. doi: 10.1007/s12032-011-9846-7. Epub 2011 Feb 8. PMID 21301998
- [Background] Coughlin SS, Calle EE, Teras LR, Petrelli J, Thun MJ. Diabetes mellitus as a predictor of cancer mortality in a large cohort of US adults. Am J Epidemiol. 2004 Jun 15;159(12):1160-7. doi: 10.1093/aje/kwh161. PMID 15191933
- [Background] Pollak M. Insulin and insulin-like growth factor signalling in neoplasia. Nat Rev Cancer. 2008 Dec;8(12):915-28. doi: 10.1038/nrc2536. PMID 19029956
- [Background] Pannala R, Basu A, Petersen GM, Chari ST. New-onset diabetes: a potential clue to the early diagnosis of pancreatic cancer. Lancet Oncol. 2009 Jan;10(1):88-95. doi: 10.1016/S1470-2045(08)70337-1. PMID 19111249
- [Background] Appleman VA, Ahronian LG, Cai J, Klimstra DS, Lewis BC. KRAS(G12D)- and BRAF(V600E)-induced transformation of murine pancreatic epithelial cells requires MEK/ERK-stimulated IGF1R signaling. Mol Cancer Res. 2012 Sep;10(9):1228-39. doi: 10.1158/1541-7786.MCR-12-0340-T. Epub 2012 Aug 7. PMID 22871572
- [Background] Schaeffer DF, Owen DR, Lim HJ, Buczkowski AK, Chung SW, Scudamore CH, Huntsman DG, Ng SS, Owen DA. Insulin-like growth factor 2 mRNA binding protein 3 (IGF2BP3) overexpression in pancreatic ductal adenocarcinoma correlates with poor survival. BMC Cancer. 2010 Feb 23;10:59. doi: 10.1186/1471-2407-10-59. PMID 20178612
- [Background] Sah RP, Nagpal SJ, Mukhopadhyay D, Chari ST. New insights into pancreatic cancer-induced paraneoplastic diabetes. Nat Rev Gastroenterol Hepatol. 2013 Jul;10(7):423-33. doi: 10.1038/nrgastro.2013.49. Epub 2013 Mar 26. PMID 23528347
- [Background] Dombrowski F, Mathieu C, Evert M. Hepatocellular neoplasms induced by low-number pancreatic islet transplants in autoimmune diabetic BB/Pfd rats. Cancer Res. 2006 Feb 1;66(3):1833-43. doi: 10.1158/0008-5472.CAN-05-2787. PMID 16452245
- [Background] Sadeghi N, Abbruzzese JL, Yeung SC, Hassan M, Li D. Metformin use is associated with better survival of diabetic patients with pancreatic cancer. Clin Cancer Res. 2012 May 15;18(10):2905-12. doi: 10.1158/1078-0432.CCR-11-2994. Epub 2012 Mar 31. PMID 22465831
- [Background] Huang X, Wullschleger S, Shpiro N, McGuire VA, Sakamoto K, Woods YL, McBurnie W, Fleming S, Alessi DR. Important role of the LKB1-AMPK pathway in suppressing tumorigenesis in PTEN-deficient mice. Biochem J. 2008 Jun 1;412(2):211-21. doi: 10.1042/BJ20080557. PMID 18387000
- [Background] Kisfalvi K, Eibl G, Sinnett-Smith J, Rozengurt E. Metformin disrupts crosstalk between G protein-coupled receptor and insulin receptor signaling systems and inhibits pancreatic cancer growth. Cancer Res. 2009 Aug 15;69(16):6539-45. doi: 10.1158/0008-5472.CAN-09-0418. PMID 19679549
- [Background] Sinnett-Smith J, Kisfalvi K, Kui R, Rozengurt E. Metformin inhibition of mTORC1 activation, DNA synthesis and proliferation in pancreatic cancer cells: dependence on glucose concentration and role of AMPK. Biochem Biophys Res Commun. 2013 Jan 4;430(1):352-7. doi: 10.1016/j.bbrc.2012.11.010. Epub 2012 Nov 15. PMID 23159620
- [Background] Kalender A, Selvaraj A, Kim SY, Gulati P, Brule S, Viollet B, Kemp BE, Bardeesy N, Dennis P, Schlager JJ, Marette A, Kozma SC, Thomas G. Metformin, independent of AMPK, inhibits mTORC1 in a rag GTPase-dependent manner. Cell Metab. 2010 May 5;11(5):390-401. doi: 10.1016/j.cmet.2010.03.014. PMID 20444419
- [Background] Ben Sahra I, Laurent K, Loubat A, Giorgetti-Peraldi S, Colosetti P, Auberger P, Tanti JF, Le Marchand-Brustel Y, Bost F. The antidiabetic drug metformin exerts an antitumoral effect in vitro and in vivo through a decrease of cyclin D1 level. Oncogene. 2008 Jun 5;27(25):3576-86. doi: 10.1038/sj.onc.1211024. Epub 2008 Jan 21. PMID 18212742
- [Background] Ben Sahra I, Regazzetti C, Robert G, Laurent K, Le Marchand-Brustel Y, Auberger P, Tanti JF, Giorgetti-Peraldi S, Bost F. Metformin, independent of AMPK, induces mTOR inhibition and cell-cycle arrest through REDD1. Cancer Res. 2011 Jul 1;71(13):4366-72. doi: 10.1158/0008-5472.CAN-10-1769. Epub 2011 May 3. PMID 21540236
- [Background] Hirsch HA, Iliopoulos D, Tsichlis PN, Struhl K. Metformin selectively targets cancer stem cells, and acts together with chemotherapy to block tumor growth and prolong remission. Cancer Res. 2009 Oct 1;69(19):7507-11. doi: 10.1158/0008-5472.CAN-09-2994. Epub 2009 Sep 14. PMID 19752085
- [Background] Lonardo E, Cioffi M, Sancho P, Sanchez-Ripoll Y, Trabulo SM, Dorado J, Balic A, Hidalgo M, Heeschen C. Metformin targets the metabolic achilles heel of human pancreatic cancer stem cells. PLoS One. 2013 Oct 18;8(10):e76518. doi: 10.1371/journal.pone.0076518. eCollection 2013. PMID 24204632
- [Background] Wang LW, Li ZS, Zou DW, Jin ZD, Gao J, Xu GM. Metformin induces apoptosis of pancreatic cancer cells. World J Gastroenterol. 2008 Dec 21;14(47):7192-8. doi: 10.3748/wjg.14.7192. PMID 19084933
- [Background] Zhuang Y, Miskimins WK. Metformin induces both caspase-dependent and poly(ADP-ribose) polymerase-dependent cell death in breast cancer cells. Mol Cancer Res. 2011 May;9(5):603-15. doi: 10.1158/1541-7786.MCR-10-0343. Epub 2011 Mar 21. PMID 21422199
- [Background] Schneider MB, Matsuzaki H, Haorah J, Ulrich A, Standop J, Ding XZ, Adrian TE, Pour PM. Prevention of pancreatic cancer induction in hamsters by metformin. Gastroenterology. 2001 Apr;120(5):1263-70. doi: 10.1053/gast.2001.23258. PMID 11266389
- [Background] Mohammed A, Janakiram NB, Brewer M, Ritchie RL, Marya A, Lightfoot S, Steele VE, Rao CV. Antidiabetic Drug Metformin Prevents Progression of Pancreatic Cancer by Targeting in Part Cancer Stem Cells and mTOR Signaling. Transl Oncol. 2013 Dec 1;6(6):649-59. doi: 10.1593/tlo.13556. eCollection 2013 Dec 1. PMID 24466367
- [Background] Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond). 2012 Mar;122(6):253-70. doi: 10.1042/CS20110386. PMID 22117616
- [Background] Owen MR, Doran E, Halestrap AP. Evidence that metformin exerts its anti-diabetic effects through inhibition of complex 1 of the mitochondrial respiratory chain. Biochem J. 2000 Jun 15;348 Pt 3(Pt 3):607-14. PMID 10839993
- [Background] El-Mir MY, Nogueira V, Fontaine E, Averet N, Rigoulet M, Leverve X. Dimethylbiguanide inhibits cell respiration via an indirect effect targeted on the respiratory chain complex I. J Biol Chem. 2000 Jan 7;275(1):223-8. doi: 10.1074/jbc.275.1.223. PMID 10617608
- [Background] Skinner HD, Crane CH, Garrett CR, Eng C, Chang GJ, Skibber JM, Rodriguez-Bigas MA, Kelly P, Sandulache VC, Delclos ME, Krishnan S, Das P. Metformin use and improved response to therapy in rectal cancer. Cancer Med. 2013 Feb;2(1):99-107. doi: 10.1002/cam4.54. Epub 2013 Feb 3. PMID 24133632
- [Background] Skinner HD, McCurdy MR, Echeverria AE, Lin SH, Welsh JW, O'Reilly MS, Hofstetter WL, Ajani JA, Komaki R, Cox JD, Sandulache VC, Myers JN, Guerrero TM. Metformin use and improved response to therapy in esophageal adenocarcinoma. Acta Oncol. 2013 Jun;52(5):1002-9. doi: 10.3109/0284186X.2012.718096. Epub 2012 Sep 5. PMID 22950385
- [Background] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Background] Niraula S, Dowling RJ, Ennis M, Chang MC, Done SJ, Hood N, Escallon J, Leong WL, McCready DR, Reedijk M, Stambolic V, Goodwin PJ. Metformin in early breast cancer: a prospective window of opportunity neoadjuvant study. Breast Cancer Res Treat. 2012 Oct;135(3):821-30. doi: 10.1007/s10549-012-2223-1. Epub 2012 Aug 30. PMID 22933030
- [Background] Dowling RJ, Niraula S, Chang MC, Done SJ, Ennis M, McCready DR, Leong WL, Escallon JM, Reedijk M, Goodwin PJ, Stambolic V. Changes in insulin receptor signaling underlie neoadjuvant metformin administration in breast cancer: a prospective window of opportunity neoadjuvant study. Breast Cancer Res. 2015 Mar 3;17(1):32. doi: 10.1186/s13058-015-0540-0. PMID 25849721
- [Background] Bonanni B, Puntoni M, Cazzaniga M, Pruneri G, Serrano D, Guerrieri-Gonzaga A, Gennari A, Trabacca MS, Galimberti V, Veronesi P, Johansson H, Aristarco V, Bassi F, Luini A, Lazzeroni M, Varricchio C, Viale G, Bruzzi P, Decensi A. Dual effect of metformin on breast cancer proliferation in a randomized presurgical trial. J Clin Oncol. 2012 Jul 20;30(21):2593-600. doi: 10.1200/JCO.2011.39.3769. Epub 2012 May 7. PMID 22564993
- [Background] Cazzaniga M, DeCensi A, Pruneri G, Puntoni M, Bottiglieri L, Varricchio C, Guerrieri-Gonzaga A, Gentilini OD, Pagani G, Dell'Orto P, Lazzeroni M, Serrano D, Viale G, Bonanni B. The effect of metformin on apoptosis in a breast cancer presurgical trial. Br J Cancer. 2013 Nov 26;109(11):2792-7. doi: 10.1038/bjc.2013.657. Epub 2013 Oct 24. PMID 24157825
- [Background] Ballehaninna UK, Chamberlain RS. The clinical utility of serum CA 19-9 in the diagnosis, prognosis and management of pancreatic adenocarcinoma: An evidence based appraisal. J Gastrointest Oncol. 2012 Jun;3(2):105-19. doi: 10.3978/j.issn.2078-6891.2011.021. PMID 22811878
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Tie J, Kinde I, Wang Y, Wong HL, Roebert J, Christie M, Tacey M, Wong R, Singh M, Karapetis CS, Desai J, Tran B, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA as an early marker of therapeutic response in patients with metastatic colorectal cancer. Ann Oncol. 2015 Aug;26(8):1715-22. doi: 10.1093/annonc/mdv177. Epub 2015 Apr 7. PMID 25851626
- [Background] Castells A, Puig P, Mora J, Boadas J, Boix L, Urgell E, Sole M, Capella G, Lluis F, Fernandez-Cruz L, Navarro S, Farre A. K-ras mutations in DNA extracted from the plasma of patients with pancreatic carcinoma: diagnostic utility and prognostic significance. J Clin Oncol. 1999 Feb;17(2):578-84. doi: 10.1200/JCO.1999.17.2.578. PMID 10080602
- [Background] Kinugasa H, Nouso K, Miyahara K, Morimoto Y, Dohi C, Tsutsumi K, Kato H, Matsubara T, Okada H, Yamamoto K. Detection of K-ras gene mutation by liquid biopsy in patients with pancreatic cancer. Cancer. 2015 Jul 1;121(13):2271-80. doi: 10.1002/cncr.29364. Epub 2015 Mar 30. PMID 25823825
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Wang Y, Chen ZE, Nikolaidis P, McCarthy RJ, Merrick L, Sternick LA, Horowitz JM, Yaghmai V, Miller FH. Diffusion-weighted magnetic resonance imaging of pancreatic adenocarcinomas: association with histopathology and tumor grade. J Magn Reson Imaging. 2011 Jan;33(1):136-42. doi: 10.1002/jmri.22414. PMID 21182131
- [Background] Niwa T, Ueno M, Ohkawa S, Yoshida T, Doiuchi T, Ito K, Inoue T. Advanced pancreatic cancer: the use of the apparent diffusion coefficient to predict response to chemotherapy. Br J Radiol. 2009 Jan;82(973):28-34. doi: 10.1259/bjr/43911400. PMID 19095814
- [Background] Cuneo KC, Chenevert TL, Ben-Josef E, Feng MU, Greenson JK, Hussain HK, Simeone DM, Schipper MJ, Anderson MA, Zalupski MM, Al-Hawary M, Galban CJ, Rehemtulla A, Feng FY, Lawrence TS, Ross BD. A pilot study of diffusion-weighted MRI in patients undergoing neoadjuvant chemoradiation for pancreatic cancer. Transl Oncol. 2014 Oct 24;7(5):644-9. doi: 10.1016/j.tranon.2014.07.005. eCollection 2014 Oct. PMID 25389460
- [Background] Blumer I, Hadar E, Hadden DR, Jovanovic L, Mestman JH, Murad MH, Yogev Y. Diabetes and pregnancy: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2013 Nov;98(11):4227-49. doi: 10.1210/jc.2013-2465. PMID 24194617
- [Background] Kurosawa J, Tawada K, Mikata R, Ishihara T, Tsuyuguchi T, Saito M, Shimofusa R, Yoshitomi H, Ohtsuka M, Miyazaki M, Yokosuka O. Prognostic relevance of apparent diffusion coefficient obtained by diffusion-weighted MRI in pancreatic cancer. J Magn Reson Imaging. 2015 Dec;42(6):1532-7. doi: 10.1002/jmri.24939. Epub 2015 May 6. PMID 25946483